CLINICAL TRIAL: NCT05455489
Title: The GIOTTO4 Study: GISE Registry of Transcatheter Treatment of Mitral Valve Regurgitation With the MitraClip G4
Brief Title: GISE Registry of Transcatheter Treatment of Mitral Valve Regurgitation With the MitraClip G4
Status: Recruiting | Type: Observational
Sponsor: Fondazione GISE Onlus (Other)
Collaborators: University of Padova (Other); Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: GISE_GIOTTO4
Record Dates: First submitted 2022-07-04; First posted 2022-07-13 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Mitral Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FUNCTIONAL MR: Patients with symptomatic severe secondary MR (3-4+, according to the multiparametric study algorithm), both ischemic or non-ischemic etiology, on optimal medical therapy
- DEGENERATIVE MR: Patients with symptomatic severe primary MR (3-4+, according to the multiparametric study algorithm)

SUMMARY:
The aim of the GISE study is to confirm the MitraClip safety and improve the device effectiveness in a selected all comers ("more-comers") population with symptomatic severe mitral regurgitation undergoing/undergone Transcatheter Edge-to-Edge Repair (TEER) with MitraClip G4.

ELIGIBILITY:
Inclusion Criteria:

SUBGROUP A: FUNCTIONAL MR Patients with symptomatic severe secondary MR (3-4+, according to the multiparametric study algorithm), both ischemic or non-ischemic etiology, on optimal medical therapy AND

* Left Ventricular End-Systolic Dimension <70 mm
* Mitral Valve area > 4 cmq
* Left ventricular ejection fraction ≥20%
* NYHA functional class II, III, ambulatory IV
* brain natriuretic peptide BNP ≥300 pg/ml or N-terminal prohormone of brain natriuretic peptide NT-proBNP ≥1500 pg/ml and/or at least one hosp for HF (Heart failure) in the 12 months prior to enrollment
* Age 18 years or older
* Subject has been adequately treated per applicable standards, including for coronary artery disease, LV (left ventricular) dysfunction, MR Mitral (regurgitation) and HF
* Local Heart-team decision SUBGROUP B: DEGENERATIVE MR Patients with symptomatic severe primary MR (3-4+, according to the multiparametric study algorithm) AND
* Mobile mitral valve (MV) length of PL ≥8 mm in case of NT device, ≥10 mm in case of XT device
* MV area > 4 cm2
* NYHA functional class > II
* Age 18 years or older
* Local HT decision In case of patients with a coexistence of both etiologies, they will be assigned to a subgroup based on the prevailing mechanism.

THE MULTIPARAMETRIC ALGORITHM FOR MR GRADING The multiparametric algorithm, adapted from the criteria recommended by the American Society of Echocardiography 2003 Guidelines and based on 3 tiers of evaluation, will be used for qualification purposes to determine if MR was 3+ or higher. The 3 tiers of evaluation are applied in a hierarchical manner (from tier 1 to 3) and patients qualified for TEER by meeting the criteria of at least one of them. For MR grading purposes, MR severity was subsequently graded as 3+ or 4+ based on the integrative evaluation of multiple parameters recommended by the The American Society of Echocardiography (ASE)

Exclusion Criteria:

* Significant right ventricular disfunction (TAPSE<15 mm and/or S'<8cm/s)
* Systolic pulmonary artery > 70 mmHg with irreversible precapillary pulmonary hypertension
* Severe TR Tricuspid valve regurgitation
* Hemodynamic instability/NYHA IV
* Impaired mobility as a result of neurological or musculoskeletal disease, or advanced dementia
* Leaflet anatomy which may preclude MitraClip implantation, proper MitraClip positioning on the leaflets or sufficient reduction in MR by the MitraClip
* Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, infiltrative cardiomyopathies
* CABG coronary artery bypass graft, PCI percutaneous coronary intervention, TAVR transcatheter aortic valve replacement, CVA cardiovascular accident within the prior 60 days
* Life expectancy <12 months due to non-cardiac conditions
* Active infections
* Advanced HF (ESC/HFA Heart Failure Association Criteria) or Bridge tp to HTx/LVAD (left ventricular assist device)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing/undergone to TEER procedure with MitraClip G4 in selected hospitals linked to the GISE network. Patients should meet all the inclusion criteria and none of the exclusion criteria; such criteria will identify a selected all comers ("more-comers") population which includes the vast majority of patients treated with MitraClip in daily practice. Retrospective enrolments are allowed if available data are in line with the study requirements and the patients can give their consent to be enrolled in the study informed consent process. Patients who don't meet one or more of the inclusion criteria or met at least one exclusion criteria are excluded from the study; however, a selected list of baseline/procedural features and follow-up data will be recorded for excluded patients.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
percentage of participants with a mitral regurgitation (MR) | at 30 days
  grade ≤1+. Two separates subgroups will be identified according to the presence of functional (FMR) or degenerative (DMR) mitral valve disease.
percentage of participants with a mitral regurgitation (MR) | at 1 year
  grade ≤1+. Two separates subgroups will be identified according to the presence of functional (FMR) or degenerative (DMR) mitral valve disease.

SECONDARY OUTCOMES:
composite of all-cause death and hospitalization for heart failure (HF), | at 30 days
  all-cause death, cardiovascular death and non-cardiovascular death, myocardial infarction, hospitalizations for HF,
composite of all-cause death and hospitalization for heart failure (HF), | at 1 year
  all-cause death, cardiovascular death and non-cardiovascular death, myocardial infarction, hospitalizations for HF,
composite of all-cause death and hospitalization for heart failure (HF), | at 2 years
  all-cause death, cardiovascular death and non-cardiovascular death, myocardial infarction, hospitalizations for HF,
composite of all-cause death and hospitalization for heart failure (HF), | at 3 years
  all-cause death, cardiovascular death and non-cardiovascular death, myocardial infarction, hospitalizations for HF,
composite of all-cause death and hospitalization for heart failure (HF), | at 4 years
  all-cause death, cardiovascular death and non-cardiovascular death, myocardial infarction, hospitalizations for HF,
composite of all-cause death and hospitalization for heart failure (HF), | at 5 years
  all-cause death, cardiovascular death and non-cardiovascular death, myocardial infarction, hospitalizations for HF,

CONTACTS AND LOCATIONS:
Locations (1):
- I.R.C.C.S. Policlinico San Donato, San Donato Milanese, Milano, Italy